CLINICAL TRIAL: NCT03133611
Title: Automatic Acoustic Speech Analysis and REM Sleep Behaviour Disorder for Detecting Subjects at High Risk for Parkinson's Disease and Other Alpha-synucleinopathies
Brief Title: Detecting Parkinson's Disease Through Speech Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Czech Technical University in Prague (Other)
Collaborators: General University Hospital, Prague (Other); University Hospital, Montpellier (Other); Mayo Clinic (Other); McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); Medical University Innsbruck (Other); San Raffaele University Hospital, Italy (Other); Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MJFF-2016-12546
Record Dates: First submitted 2017-04-26; First posted 2017-04-28 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Parkinson Disease; REM Sleep Behavior Disorder
Keywords: Speech disorder; Acoustic analysis; Dysarthria
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder; Speech Disorders; Dysarthria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parkinson's disease (Other): Speech assessment. Routine clinical assessment.
  Interventions: Other: Speech assessment; Other: Routine clinical assessment
- REM sleep behaviour disorder (Other): Speech assessment. Routine clinical assessment.
  Interventions: Other: Speech assessment; Other: Routine clinical assessment
- Healthy controls (Other): Speech assessment. Routine clinical assessment.
  Interventions: Other: Speech assessment; Other: Routine clinical assessment

INTERVENTIONS:
Other: Speech assessment — Each subject will undergo short non-invasive speech assessment lasting approximately 15 minutes that will be recorded using microphone.
Other: Routine clinical assessment — Volunteers who enroll in the study will undergo various assessments lasting about 2 hours, including neurological examination of both motor and non-motor skills, autonomic testing and cognitive testing.

SUMMARY:
Speech is an important indicator of motor function and movement coordination and can be extremely sensitive to involvement in the course of neurologic diseases. The aim of this project is to discover for the first time using simple speech recording and high end pattern analysis preclinical stages of disabling central nervous system disorders including Parkinson's disease and other alpha-synucleinopathies in "at high risk" patients with REM sleep behavior disorder and thus provide one essential prerequisite for trials on REM sleep behavior disorder with preventive therapy.

DETAILED DESCRIPTION:
Seven centers of excellence in sleep research will investigate speech and other clinical symptoms in more than 100 subjects with REM sleep behavior disorder. Analyses of a number of unique speech dimensions based upon three fundamental categories of simple speaking tasks will be used to search for specific prodromal alterations in speech patterns in REM sleep behavior disorder, compared to age- and gender-matched patients with early Parkinson's disease and healthy control subjects. Robust algorithms allowing automated speech analysis will be developed and optimized through English, German, French, Czech and Italian languages. Early motor dysfunction strongly predicts Parkinson's disease and other alpha-synucleinopathies. In this regard, vocal assessment has intriguing potential advances as is non-invasive, inexpensive, simple to administer and scalable to large population with possibility to perform recordings remotely, even by telephone from patients' home. Speech analysis may serve as a simple tool to screen large populations for the risk to develop Parkinson's disease. If speech impairment appears to be a strong biomarker of early motor dysfunction, the screening of speech changes may improve stratification for future neuroprotective therapies for Parkinson's disease and other synucleinopathies.

ELIGIBILITY:
Inclusion Criteria for subjects with Parkinson's disease (PD):

* Diagnosed based on the MDS Clinical Diagnostic Criteria for Parkinson's Disease including the presence of bradykinesia in combination with either rest tremor, rigidity, or both;
* Hoehn & Yahr stage 1-2 in the defined OFF state;
* Disease duration from diagnosis < 5 years;
* No motor fluctuations or dyskinesias;
* On stable dose of medication in last four weeks;
* Onset of PD after 50 years;
* No history of communication or neurological disorders unrelated to PD;
* Not currently involved in any speech therapy;

Inclusion Criteria for subjects with REM Sleep Behaviour Disorder (RBD):

* Fulfill criteria for RBD based on polysomnography according to the standard International Classification of Sleep Disorders diagnostic criteria, 3rd edition;
* Onset of RBD after 50 years;
* No history of communication or neurological disorders.

Inclusion Criteria for healthy control subjects:

* No history of communication or neurological disorders, parasomnias and other sleep disorders with important severity;
* No regular benzodiazepines, hypnotics and melatonin intake.

Exclusion criteria:

(for all the arms) Inability to speak and read a text aloud.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Motor Speech Disorder Examination (MSDE) | Within one session (15 minutes)
  Quantitative acoustic assessment of several deviant speech dimensions connected with phonatory, articulatory, and prosodic abnormalities in hypokinetic dysarthria of Parkinson's disease.

SECONDARY OUTCOMES:
MDS Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Within one session (30 minutes)
  The most commonly used scale for the clinical evaluation of Parkinson's disease assessing variety of motor and non-motor symptoms.
SCOPA-AUT | Within one session (30 minutes)
  Scale for assessment of autonomic dysfunction in Parkinson's disease.
Montreal Cognitive Assessment (MoCA) | Within one session (15 minutes)
  Scale for assessment of several cognitive domains.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Rusz, PhD, Study Director — Czech Technical University in Prague
Locations (7):
- Mayo Clinic, Rochester, Minnesota, United States
- Medical University of Innsbruck, Innsbruck, Austria
- McGill University Health Centre, Montreal, Quebec, Canada
- General University Hospital, Prague, CZ, Czechia
- Gui-de-Chauliac Hospital, Montpellier, France
- University of Marburg, Marburg, Hesse, Germany
- San Raffaele Hospital, Milan, Italia, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical data (speech recordings and associated clinical scales) may be shared with the Michael J. Fox Foundation (the study funder). This data may be kept for storage at a central repository either hosted by the Michael J. Fox Foundation, its collaborators, or consultants.

REFERENCES:
- [Background] Rusz J, Hlavnicka J, Tykalova T, Buskova J, Ulmanova O, Ruzicka E, Sonka K. Quantitative assessment of motor speech abnormalities in idiopathic rapid eye movement sleep behaviour disorder. Sleep Med. 2016 Mar;19:141-7. doi: 10.1016/j.sleep.2015.07.030. Epub 2015 Sep 14. PMID 26459688
- [Background] Postuma RB, Lang AE, Gagnon JF, Pelletier A, Montplaisir JY. How does parkinsonism start? Prodromal parkinsonism motor changes in idiopathic REM sleep behaviour disorder. Brain. 2012 Jun;135(Pt 6):1860-70. doi: 10.1093/brain/aws093. Epub 2012 May 4. PMID 22561644
- See also: Fox Trial Finder — https://foxtrialfinder.michaeljfox.org/trial/4937/
- See also: Michael J. Fox Foundation — https://www.michaeljfox.org/foundation/grant-detail.php?grant_id=1616